CLINICAL TRIAL: NCT00004891
Title: Prospective Evaluation of 18F-Fluorodeoxyglucose Positron Emission Tomography (FDG-PET) in the Multimodality Management of Locally Advanced Primary Rectal Cancer
Brief Title: PET and CT Scans in Patients With Locally Advanced Primary Rectal Cancer That Can Be Removed During Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MSKCC-99048; CDR0000067567 (Registry Identifier: PDQ (Physician Data Query)); NCI-G00-1695
Record Dates: First submitted 2000-03-07; First posted 2003-01-27 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Colorectal Cancer
Keywords: stage II rectal cancer; stage III rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — Drug Therapy; Neoadjuvant Therapy; Magnetic Resonance Spectroscopy; Fluorodeoxyglucose F18; Radiotherapy

ARMS (1):
- primary resectable rectal cancer (Experimental)
  Interventions: Drug: chemotherapy; Procedure: computed tomography; Procedure: conventional surgery; Procedure: neoadjuvant therapy; Procedure: positron emission tomography; Procedure: radionuclide imaging; Radiation: fludeoxyglucose F 18; Radiation: radiation therapy

INTERVENTIONS:
Drug: chemotherapy
Procedure: computed tomography
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Procedure: positron emission tomography
Procedure: radionuclide imaging
Radiation: fludeoxyglucose F 18
Radiation: radiation therapy

SUMMARY:
RATIONALE: Diagnostic procedures, such as PET and CT scans, may improve the ability to detect the extent of locally advanced primary rectal cancer and may also help to measure a patient's response to treatment.

PURPOSE: This clinical trial is studying how well PET and CT scans detect residual or metastatic disease in patients with locally advanced primary rectal cancer that can be removed during surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine if fludeoxyglucose F 18 positron emission tomography (FDG-PET) is superior to CT scan at monitoring rectal cancer response to radiation and chemotherapy by identifying residual rectal cancer in the rectal wall or pelvic lymph nodes in order to optimize selection of patients suitable for a sphincter preserving rectal cancer resection or a local excision.
* Determine the accuracy of FDG-PET in detecting extrapelvic metastatic disease in primary rectal cancer patients considered operable on the basis of currently accepted diagnostic work-up, including abdominal CT scan and chest x-ray.

OUTLINE: This is a diagnostic study conducted concurrently with multimodality management.

Within 1-2 weeks prior to starting preoperative radiotherapy/chemotherapy, patients undergo baseline positron emission tomography (PET) imaging of the thorax, abdomen, and pelvis. Patients receive fludeoxyglucose F 18 (FDG) IV followed 45 minutes later by PET imaging. Patients also undergo baseline CT imaging of the abdomen and pelvis. A CT scan of the chest is obtained if the prestudy chest x-ray is abnormal.

Patients receive preoperative radiotherapy/chemotherapy. Within 4-6 weeks of completion of radiotherapy/chemotherapy, patients undergo repeat FDG-PET imaging and CT scan. Patients undergo surgical resection 1-2 weeks later.

PROJECTED ACCRUAL: A total of 125 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Primary resectable rectal cancer as determined by currently accepted diagnostic work-up, including CT scan and endorectal ultrasound (EUS)
* Must meet criteria for preoperative radiotherapy and chemotherapy:

  * Bulky tumors and/or EUS evidence of T3-4 and/or N1 disease

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* Not pregnant or nursing
* No uncontrolled diabetes mellitus (i.e., greater than 175 mg/dL)
* No intolerance of being inside PET scanner for duration of study
* No vulnerable patients (e.g., mentally retarded or prisoners)

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics

Surgery:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 1999-09; Primary Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Determine if fludeoxyglucose F 18 positron emission tomography (FDG-PET) is superior to CT scan | 2 years
  at monitoring rectal cancer response to radiation and chemotherapy by identifying residual rectal cancer in the rectal wall or pelvic lymph nodes in order to optimize selection of patients suitable for a sphincter preserving rectal cancer resection or a local excision

SECONDARY OUTCOMES:
Determine the accuracy of FDG-PET | 2 years
  in detecting extrapelvic metastatic disease in primary rectal cancer patients considered operable on the basis of currently accepted diagnostic work-up, including abdominal CT scan and chest x-ray.

CONTACTS AND LOCATIONS:
Overall Officials: Jose G. Guillem, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Nahas CS, Akhurst T, Yeung H, Leibold T, Riedel E, Markowitz AJ, Minsky BD, Paty PB, Weiser MR, Temple LK, Wong WD, Larson SM, Guillem JG. Positron emission tomography detection of distant metastatic or synchronous disease in patients with locally advanced rectal cancer receiving preoperative chemoradiation. Ann Surg Oncol. 2008 Mar;15(3):704-11. doi: 10.1245/s10434-007-9626-y. Epub 2007 Sep 20. PMID 17882490
- [Result] Guillem JG, Puig-La Calle J Jr, Akhurst T, Tickoo S, Ruo L, Minsky BD, Gollub MJ, Klimstra DS, Mazumdar M, Paty PB, Macapinlac H, Yeung H, Saltz L, Finn RD, Erdi Y, Humm J, Cohen AM, Larson S. Prospective assessment of primary rectal cancer response to preoperative radiation and chemotherapy using 18-fluorodeoxyglucose positron emission tomography. Dis Colon Rectum. 2000 Jan;43(1):18-24. doi: 10.1007/BF02237238. PMID 10813118
- [Derived] Guillem JG, Ruby JA, Leibold T, Akhurst TJ, Yeung HW, Gollub MJ, Ginsberg MS, Shia J, Suriawinata AA, Riedel ER, Mazumdar M, Saltz LB, Minsky BD, Nash GM, Paty PB, Temple LK, Weiser MR, Larson SM. Neither FDG-PET Nor CT can distinguish between a pathological complete response and an incomplete response after neoadjuvant chemoradiation in locally advanced rectal cancer: a prospective study. Ann Surg. 2013 Aug;258(2):289-95. doi: 10.1097/SLA.0b013e318277b625. PMID 23187748